CLINICAL TRIAL: NCT06200831
Title: Simultaneous vs. Staged Resection of Colorectal Cancer With Synchronous Liver Metastases - A Multicentre Randomized Controlled Trial
Brief Title: Simultaneous vs. Staged Resection of Colorectal Cancer With Synchronous Liver Metastases
Acronym: SYLMET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other); Haukeland University Hospital (Other); St. Olavs Hospital (Other); Helse Stavanger HF (Other Government); University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Sheraz Yaqub, Principal Investigator, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201644
Record Dates: First submitted 2023-12-13; First posted 2024-01-11 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Colorectal Cancer; Colorectal Neoplasms Malignant; Liver Metastasis Colon Cancer; Liver Metastases
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Staged resection (Active Comparator): Resection of the primary colorectal carcinoma and liver metastases in two separate surgeries.
  Interventions: Procedure: Staged resection
- Simultaneous resection (Experimental): Resection of both the primary colorectal carcinoma and the liver metastases in one surgical procedure.
  Interventions: Procedure: Simultaneous resection

INTERVENTIONS:
Procedure: Staged resection — Patients randomized to staged resection will be operated according to the decision made by the tumor board meeting (liver or colorectal cancer first, based on tumor burden and symptoms), but both resections have to be done within a time period of 4-12 weeks.
  Other Names: Two-staged resection; Sequential resection
  Arms: Staged resection
Procedure: Simultaneous resection — In cases with simultaneous surgery, the liver resection is performed prior to colon resection in order to keep a low central venous pressure during the first part of the surgical procedure and to avoid congestion of the anastomosis line owing to possible Pringle manoeuvre.
  Other Names: Combined resection; Synchronous resection
  Arms: Simultaneous resection

SUMMARY:
The SYLMET Trial is a randomized trial to compare simultaneous and two-staged resection of primary colorectal and synchronous liver metastases. This is an investigator-initiated, multicentre, randomized controlled trial to assess complications (primary endpoint), survival, cost-effectiveness, and quality of life (secondary endpoints).This trial will include patients with resectable primary tumour in the colon or upper rectum with less than five liver metastases that is possible to treat with surgical resection and/or ablation (RFA/MWA) at time of evaluation.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) represents the second most common cause of cancer and cancer death in Norway, and the incidence is increasing (Cancer in Norway, 2021, Cancer Registry of Norway). The liver is the most common site of metastasis from CRC. More than 4500 individuals are diagnosed with CRC in Norway each year, and approximately 20% of patients present with liver metastases at time of diagnosis (synchronous metastases). Resection of both the primary tumor and liver metastases is considered the only curative treatment, and has been shown to improve long-term survival, and is considered standard of care. However, the optimal timing of surgical resection of synchronous liver metastases in relation to the primary tumor is not well defined. Traditionally, staged resection has been preferred (i.e., resection of the primary tumour and liver metastases on separate admissions with a period of recovery between the two operations), whereas simultaneous resection is appealing (i.e., resection of both primary and metastases in one operative session). Despite a lack of randomized controlled trials comparing these two surgical approaches, the number of simultaneous resections has increased at several institutions. The evolvement of both liver and colorectal surgery in the last decades has led to reduced complications, making simultaneous resections more feasible. Previous retrospective cohort studies and meta-analyses suggest that simultaneous and staged approach carry similar postoperative complication and perioperative mortality rates as well as long-term survival. A recently published prospective observational study on staged or simultaneous surgery, reported similar outcomes in selected patients. To date, there is only one published randomized controlled trial which was aborted after inclusion of half of the sample size, after an accrual time of 10 years18. Due to lack of evidence, the majority of surgical societies worldwide still treats this patient group with staged resections, resulting in two hospital admissions, two rounds of general anaesthesia and surgery, and finally two episodes of postoperative recovery and rehabilitation. If this trial demonstrates that simultaneous surgery is safe, feasible, and cost-effective, it will potentially have a practice-changing impact worldwide.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years old.
* Both CRC and liver metastases in situ at time of evaluation.
* Resectable primary tumor in the colon or upper rectum.
* Less than 5 liver metastases, evaluated by the multidisciplinary tumor board meeting as possible to treat with surgical resection and/or ablation (RFA/MWA).

Exclusion Criteria:

* Unresectable primary tumor.
* Locally advanced primary tumor (T4).
* Primary tumor in the lower rectum with indication for abdominoperineal resection.
* Acute or imminent bowel obstruction.
* Perforation or major bleeding from the primary tumor.
* Pre-treatment of the primary tumor with a colon stent.
* Liver resection requiring resection of more than 2 adjacent segments (Couinaud).
* Liver metastases planned treated with irreversible electroporation (IRE).
* Non-resectable lung metastases.
* Metastases outside of liver (besides resectable lung metastases).
* Eastern Cooperative Oncology Group (ECOG) Performance status ≥ 3.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Comprehensive Complication Index, CCI | 90 days
  The CCI is calculated as the sum of all complications that are weighted for their severity (multiplication of the median reference values from patients and physicians). The final formula yields a continuous scale to rank the severity of any combination of complications from 0 to 100 in a single patient.

SECONDARY OUTCOMES:
Health Economics | 1 year
  Cost-effectiveness calculated by incremental cost effectiveness ratio (ICER)
Overall survival | 3 and 5 years
  Survival
Clavien Dindo Complications | 90 days
  Scale from 1 to 5. Higher score meaning more severe complication.
Quality of Life: EQ-5D | Pre-operative, 30-days, 90-days, 6 months, 12 months
  EQ-5D is an instrument which evaluates the generic quality of life developed in Europe and widely used. The EQ-5D descriptive system is a preference-based HRQL measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The scale range from -0.224 to 1; with 0, 1, and negative values corresponding to death, full health, and health states worse than death, respectively.
Quality of Life: EORTC QLQ-30 | Pre-operative, 30-days, 90-days, 6 months, 12 months
  The EORTC Core Quality of Life questionnaire (EORTC QLQ-C30) is designed to measure cancer patients' physical, psychological and social functions. The questionnaire is composed of multi-item scales and single items. Score from 1-100.

CONTACTS AND LOCATIONS:
Overall Officials: Sheraz Yaqub, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kleive D, Aas E, Angelsen JH, Bringeland EA, Nesbakken A, Nymo LS, Schultz JK, Soreide K, Yaqub S. Simultaneous Resection of Primary Colorectal Cancer and Synchronous Liver Metastases: Contemporary Practice, Evidence and Knowledge Gaps. Oncol Ther. 2021 Jun;9(1):111-120. doi: 10.1007/s40487-021-00148-2. Epub 2021 Mar 23. PMID 33759076
- [Background] Siriwardena AK, Serrablo A, Fretland AA, Wigmore SJ, Ramia-Angel JM, Malik HZ, Stattner S, Soreide K, Zmora O, Meijerink M, Kartalis N, Lesurtel M, Verhoef C, Balakrishnan A, Gruenberger T, Jonas E, Devar J, Jamdar S, Jones R, Hilal MA, Andersson B, Boudjema K, Mullamitha S, Stassen L, Dasari BVM, Frampton AE, Aldrighetti L, Pellino G, Buchwald P, Gurses B, Wasserberg N, Gruenberger B, Spiers HVM, Jarnagin W, Vauthey JN, Kokudo N, Tejpar S, Valdivieso A, Adam R; Joint E-AHPBA/ESSO/ESCP/ESGAR/CIRSE 2022 Consensus on colorectal cancer with synchronous liver metastases. The multi-societal European consensus on the terminology, diagnosis and management of patients with synchronous colorectal cancer and liver metastases: an E-AHPBA consensus in partnership with ESSO, ESCP, ESGAR, and CIRSE. HPB (Oxford). 2023 Sep;25(9):985-999. doi: 10.1016/j.hpb.2023.05.360. Epub 2023 Jul 13. PMID 37471055
- [Background] Yaqub S, Margonis GA, Soreide K. Staged or Simultaneous Surgery for Colon or Rectal Cancer with Synchronous Liver Metastases: Implications for Study Design and Clinical Endpoints. Cancers (Basel). 2023 Apr 6;15(7):2177. doi: 10.3390/cancers15072177. PMID 37046837